CLINICAL TRIAL: NCT04760509
Title: Short- Term Follow up Of Neonates Born With Neural Tube Defect
Acronym: STFUONBWNTD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Umit Ayse Tandircioglu, Medical Doctor, Hacettepe University
Other Study IDs: GO201150
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Neural Tube Defects; Newborn Morbidity
Keywords: newborn; neural tube defects; meningomyelosel
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: In this study, the short-term follow-up of patients with neural tube defects in the neonatal intensive care unit will be evaluated retrospectively. — there is no intervention. It is retrospective study.
  Other Names: meningomyelosel

SUMMARY:
Neural tube defects (NTD), which is the most common anomaly of the central nervous system, which can be diagnosed during antenatal period, brings many problems both in the neonatal period and in advanced ages. Open neural tube defects, in particular, progress with sensory-motor deficits due to the risk of infection and neural tissue loss from birth, and should be followed closely from the neonatal period. Newborns born with a neural tube defect should be operated within the first 72 hours postnatal and the defect should be closed.

In this hospital, newborns with NTD are monitored in our neonatal surgery intensive care unit before and after surgery. Neonatal specialists, neurosurgeons and other specialists when there is an additional anomaly evaluate the baby as multidisciplinary.

In this project, the short-term follow-up data of babies with NTD who have been followed up in this neonatal surgery intensive care unit for the last fifteen years will be evaluated retrospectively.

DETAILED DESCRIPTION:
Neural tube defects (NTD), which is the most common anomaly of the central nervous system, which can be diagnosed during antenatal period, brings many problems both in the neonatal period and in advanced ages. Open neural tube defects, in particular, progress with sensory-motor deficits due to the risk of infection and neural tissue loss from birth, and should be followed closely from the neonatal period. Newborns born with a neural tube defect should be operated within the first 72 hours postnatal and the defect should be closed.

In this hospital, newborns with NTD are monitored in neonatal surgery intensive care unit before and after surgery. Neonatal specialists, neurosurgeons and other specialists when there is an additional anomaly evaluate the baby as multidisciplinary.

In this project, the short-term follow-up data of babies with NTD who have been followed up in neonatal surgery intensive care unit for the last fifteen years will be evaluated retrospectively.Information of patients hospitalized with a diagnosis of neural tube defect in the neonatal intensive care unit between January 1, 2006 and January 1, 2021 will be recorded in the file. In addition to demographic information such as antenatal follow-up data of patients, maternal diseases, birth weights, birth weeks, delivery types, neurological examinations, laboratory findings, imaging (such as graphy, tomography, ultrasonography), surgery notes, additional anomalies from the hospital system retrospectively will be saved. Immediately after babies with NTD are born, the defect should be protected in the delivery room with a wet sterile sponge and the baby should be placed in a lateral or prone position. Since the risk of meningitis is high and the destruction of the neural tissue within the pouch will increase within days, the sac repair should be performed within the first 72 hours. Antibiotics should be initiated empirically in these patients with high risk of meningitis. In the postoperative follow-up; The patient should be monitored in terms of wound infection of the repaired sac, bosom leakage, fistula formation and hydrocephalus.

In this study, the short-term follow-up of patients with neural tube defects in the neonatal intensive care unit will be evaluated retrospectively. As a result of this data evaluation to be made over the hospital information system, "Hacettepe University Neonatal Intensive Care Unit patient follow-up with NTD" will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Babies who have been hospitalized in the Neonatal Intensive Care Unit of Hacettepe University İhsan Dogramaci Children's Hospital and who have been operated due to neural tube defects will be taken.

Exclusion Criteria:

* Patients whose file records cannot be reached will not be included.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The method and data collection tools of the study: the information of the patients hospitalized in the neonatal intensive care unit with a diagnosis of neural tube defect between January 1, 2006 and January 1, 2021 will be recorded in the file. In addition to demographic information such as antenatal follow-up data, maternal diseases, birth weights, birth weeks, delivery types of patients, neurological examinations, laboratory findings, imaging (such as graphy, tomography, ultrasonography), surgery during the follow-up in our unit.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the day of surgery to be performed in the postnatal period | 8 months
  It is aimed to demonstrate the effects of early or late surgery day on the baby in the postnatal period.

CONTACTS AND LOCATIONS:
Locations (1):
- Umit Ayse Tandircioglu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The method and data collection tools of the study: The committee, the information of the patients hospitalized in the neonatal intensive care unit with a diagnosis of neural tube defect between January 1, 2006 and January 1, 2021 will be recorded in the file. In addition to demographic information such as antenatal follow-up data, maternal diseases, birth weights, birth weeks, delivery types of patients, neurological examinations, laboratory findings, imaging (such as graphy, tomography, ultrasonography), surgery during the follow-up in our unit.

REFERENCES:
- [Background] Richard J. Martin, MBBS, FRACP, Avroy A. Fanaroff, MD, FRCPE, FRCPCH, Michele C. Walsh, MD, MSE Fanaroff and Martin's Neonatal-Perinatal Medicine. Diseases of the Fetus and Infant. 11th Edition 1073- 1080.
- [Result] McLone DG. Care of the neonate with a myelomeningocele. Neurosurg Clin N Am. 1998 Jan;9(1):111-20. PMID 9405769